CLINICAL TRIAL: NCT06633237
Title: Effectiveness of Core Training on the Biomechanics of Jump Landing in Amateur Female Basketball Players: a Cluster Randomized Controlled Trial
Brief Title: Effectiveness of Core Training on the Biomechanics of Jump Landing in Amateur Female Basketball Players
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Eduard Mercader Vila, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FIS-2023-10
Record Dates: First submitted 2024-10-05; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Landing Biomechanics; Jumping Performance; Trunk Stability
Keywords: Core training; Jump-landing biomechanics; Jump performance; Female basketball players; Landing Error Scoring System (LESS); Trunk stability; Amateur athletes; Injury prevention

STUDY DESIGN:
Intervention Model Description: Cluster parallel randomized clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core training program (Experimental): This group will participate in the core training intervention integrated into the warm-up during basketball training sessions. The core training program will be applied twice a week for 8 weeks. The intervention focuses on improving core and trunk stability to reduce jump-landing errors and enhance jumping performance.
  Interventions: Other: Core training program in female amateur basketball players
- Standard warm-up (No Intervention): This group will participate in the core training intervention integrated into the warm-up during basketball training sessions. The core training program will be applied twice a week for 8 weeks. The intervention focuses on improving core and trunk stability to reduce jump-landing errors and enhance jumping performance.

INTERVENTIONS:
Other: Core training program in female amateur basketball players — The intervention consists of a core training program specifically designed to improve core and trunk stability in female amateur basketball players. The program is integrated into the warm-up routine and is applied twice a week over an 8-week period. Each session lasts approximately 12-15 minutes and includes five exercises. The training program is divided into three phases of progression, gradually increasing the difficulty of the exercises over the 8 weeks by incorporating more dynamic and functional movements.
  Other Names: Core training program in female amateur basketball players 2024
  Arms: Core training program

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a core training intervention on jump-landing biomechanics in female amateur basketball players. Additionally, it will assess the impact of this intervention on jumping performance. The primary questions it aims to answer are:

1. Does a core training intervention reduce jump-landing biomechanics errors, as measured by the Landing Error Scoring System (LESS)?
2. Will the LESS items related to core and trunk stability improve following the core training program?
3. Will the core training program enhance jumping performance in female amateur basketball players?
4. Is there a relationship between poor LESS scoring and poor jumping performance? Researchers will compare the effects of a core training intervention applied during the warm-up in basketball training with the standard warm-up routine typically used at this basketball level.

Participants will be asked to:

* Attend the scheduled assessments at three points during the study: before the intervention begins, at the end of the 8-week intervention period, and after a 3-month follow-up period.
* Teams in the intervention group will incorporate the core training exercises during their warm-up, twice a week, over the 8-week period.
* Teams in the control group will continue their standard warm-up routine without any modifications.
* All participating teams will document the training sessions completed by the players to monitor adherence to the program.

DETAILED DESCRIPTION:
This clinical trial aims to evaluate the effectiveness of a core training intervention on jump-landing biomechanics and jumping performance in female amateur basketball players. Given the high incidence of lower limb injuries in this population, it is essential to identify training interventions that can reduce injury risk and enhance athletic performance.

This is a cluster parallel randomized clinical trial involving female amateur basketball teams. Participants will be randomly assigned to either the intervention group, which will receive core training during warm-up sessions, or the control group, which will continue with their standard warm-up.

The primary objectives of this study are to:

* To investigate the effect of a core training program on biomechanical alterations, measured using the Landing Error Scoring System (LESS), during jump landings in female amateur basketball players.
* To analyze the results of LESS items in a sample of female amateur basketball players.

The secondary objectives are to:

* To examine the effect of a core training program on jumping performance in female amateur basketball players.
* To identify associations between LESS results and jumping performance among female amateur basketball players.

Intervention: The core training program is designed to improve core and trunk stability and is incorporated into the warm-up routine. The program will consist of two sessions per week over an 8-week period, with each session lasting approximately 12-15 minutes. Each session will include five core exercises that will be progressively more challenging across three phases throughout the 8 weeks, integrating dynamic and functional movements.

Participants: Eligible participants will be female amateur basketball players who are actively registered and federated with the Catalan Basketball Federation at the time of the study. All players will have undergone an annual medical examination to ensure they are healthy athletes. Participation will be voluntary, and all participants must sign an informed consent form. In the case of minors, the legal guardian will be informed and must consent to their participation by signing the informed consent form.

If a player is excluded from participation in the study or chooses not to participate, no tests or data collection will be conducted on that athlete. However, they will continue with their team's established warm-up program, whether it is the standard program (control group) or the protocolized core training program (intervention group). The warm-up routines for both groups are standard practices and will be implemented by the team coaches for the entire team to facilitate logistics during training sessions. It is deemed impractical to apply the program individually to the participants in the study, and the implementation of a warm-up protocol does not significantly alter the training dynamics of the team.

Assessments: Assessments will take place at the sports facilities of the participating teams on the same day for all team members. Before the evaluations, participants will be asked to perform a minimum of 5 minutes of free warm-up to prepare for the tests.

Data Collection:

Initial Questionnaire: At the beginning of the study, each participant will complete a questionnaire that includes information about:

* Age
* Height
* Weight
* Injury history
* Age of menarche
* Other sports activities participated in
* Years of practice in basketball Only the participants' email addresses will be collected to relate it to the assessments, without gathering any other personal data.

Jump Testing:

Participants will perform three jump tests (Drop Vertical Jump, DVJ), which will be filmed for later evaluation. The reception of these jumps will take place on the Chronojump contact platform to capture the results regarding vertical jump height. The jump analysis will be recorded simultaneously from frontal and lateral positions, using two smartphones set to 60 frames per second (FPS). The phones will be placed 3.5 m away from the jump platform and at a height of 1.20 m from the ground. The jump achieving the maximum height will be selected for analysis, and the video corresponding to this jump will be used for the LESS evaluation.

Results Analysis:

Data from the study will be collected in a spreadsheet and managed using the Jamovi statistical analysis software. The results from the LESS evaluation will be described as follows:

* A description of the overall LESS score will be provided, using either mean and standard deviation (SD) or median and interquartile range (IQR), depending on data distribution. This description will be made for each sports category.
* Frequencies and percentages for the presence of errors in each LESS category will be presented, with the exception of items 16 and 17, which address general aspects and do not provide specific information on biomechanical alterations.

To evaluate the effect of the core training program on LESS scores and vertical jump performance during the DVJ, the following analyses will be performed:

* A repeated measures ANOVA will be used to determine if there are changes over time within the same group (intervention or control) across different time points. A post-hoc analysis will follow to identify at which time points (T0, T1, and T2) these changes occur. If the data does not follow a normal distribution, the Friedman test will be applied.
* For between-group comparisons (control and intervention) at different time points (T0, T1, and T2), a Student's T-test will be performed if the data is normally distributed. If the data does not follow normality, the Mann-Whitney U test will be used.
* Subgroup analyses will be conducted for each sports category, as well as for a subgroup with a history of lower limb injuries. Participants will be considered to have a history of injury if they have undergone surgery on a lower limb or have had an injury resulting in more than 3 months of sports inactivity in the last two sports seasons.

To identify associations between LESS results and jump performance, a Pearson correlation analysis will be performed between the LESS score and the vertical jump height during the DVJ. The following correlation thresholds will be used:

R < 0.10 → No correlation R ≥ 0.10 and < 0.30 → Small correlation R ≥ 0.30 and < 0.50 → Moderate correlation R ≥ 0.50 → Strong correlation The significance level for the study will be set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Be a licensed player and part of the official roster of a participating team.
* Be at least 13 years old at the time of the study.
* Have reached menarche prior to the start of the study.
* Be actively training and competing regularly at the time of the study.
* Have completed at least one full competitive season prior to the start of the study.

Exclusion Criteria:

* Have an injury or illness at the time of the study that prevents proper participation in the assessments.
* Sustain an injury during the intervention period that affects participation.
* Failure to complete at least 80% of the prescribed program.
* Be absent during any of the scheduled assessment sessions.

Min Age: 13 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the mean Landing Error Scoring System (LESS) score after 8-week intervention and 3-month follow-up | From baseline (pre-intervention), after 8 weeks of intervention, and at 3-month follow-up.
  The primary outcome measure is the change in the mean score of the Landing Error Scoring System (LESS) at three time points: baseline (pre-intervention), immediately after the 8-week intervention, and following a 3-month follow-up period. The LESS is a validated observational tool used to assess jump-landing biomechanics, focusing on errors in movement patterns that may increase injury risk. Participants will perform a Drop Vertical Jump (DVJ) task, which will be recorded and analyzed. A single trained evaluator will assess the video recordings using the LESS criteria. A lower LESS score indicates fewer movement errors and improved jump-landing biomechanics.

SECONDARY OUTCOMES:
Change in jump height measured during drop vertical jump (DVJ) using a contact platform | From baseline (pre-intervention), after 8 weeks of intervention, and at 3-month follow-up.
  The secondary outcome measure is the change in jump height during the Drop Vertical Jump (DVJ), assessed using a Chronojump contact platform (Boscosystem). Participants will perform a DVJ by jumping from a 30 cm box to a horizontal distance equivalent to 50% of their height. Each participant will complete three valid jumps, and the data collected will be the maximum height achieved across these three jumps. The jump will be followed by a landing on the Chronojump platform, which will record the maximum jump height achieved. This assessment will be performed at three time points: baseline (pre-intervention), immediately after the 8-week intervention, and at a 3-month follow-up. A higher jump height indicates improved jumping performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No